CLINICAL TRIAL: NCT05971017
Title: Evaluation of Potential Health Effects of Biostimulated Lettuce for Human Population
Brief Title: Health Effects of Biostimulated Lettuce in Human
Acronym: NUTRIWEED23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sara Baldassano, PROFESSOR, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Weed2023
Record Dates: First submitted 2023-07-12; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Nutrition, Healthy; Dietary Deficiency; Bone Resorption; Glucose Metabolism Disorders; Lipid Metabolism Disorder; Hepatic Steatosis
MeSH Terms: conditions — Malnutrition; Bone Resorption; Glucose Metabolism Disorders; Lipid Metabolism Disorders; Fatty Liver | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: control group, biostimulated group
Who Masked: Participant
Masking Description: Two groups that consumed lettuce. No differences in shape, size, colours of lettuce
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): To the control group was assigned lettuce without any biostimulation but with the same characteristic of biostimulated lettuce (soil, water, harvesting time)
  Interventions: Dietary Supplement: Control Group
- Biostimulated Group (Experimental): experimental: Biostimulated group: To the intervention group was assigned the biostimulated lettuce.
  Interventions: Dietary Supplement: Biostimulated group

INTERVENTIONS:
Dietary Supplement: Control Group — Lettuce without any biostimulation was assigned to each participant belonging to the control group which ate 100gr every day for 15 days
  Other Names: Placebo Comparator
  Arms: Control group
Dietary Supplement: Biostimulated group — Intervention biostimulated group 100gr of biostimulated lettuce were assigned to each participant belonging to the intervention group which ate 100 grams every day for a total of 15 days
  Other Names: Intervention group
  Arms: Biostimulated Group

SUMMARY:
The aim of the project is to study the influence of biostimulate crops on a healthy population in order to assess influence on hematological parameters and specific metabolism (glucose, lipid, iron, bone) and gut and lipid hormones. Secondary outcome will be to find out micronutrient presence in urine and serum. The use of biostimulation in modern agriculture has rapidly expanded in recent years, owing to their beneficial effects on crop yield and product quality, which have come under the scope of intensive research.

DETAILED DESCRIPTION:
The aim of the project is to study the influence of biostimulated crops on a healthy population in order to assess influence on hematological parameters and specific metabolism (glucose, lipid, iron, bone) and gut and lipid hormones. Secondary outcome will be to find out micronutrient presence in urine and serum in order to evaluate vegetables as carrier. The use of biostimulation in modern agriculture has rapidly expanded in recent years, owing to their beneficial effects on crop yield and product quality, which have come under the scope of intensive research.

The present project aims to investigate the benefits of biostimulated lettuce in a cohort of healthy individuals. For biostimulation are used organic and inorganic compounds or microorganisms that when applied to plants can enhance plants' growth, yield, and tolerance to stress. Participants will be fed with differently biostimulated lettuces to study the influence on hematological parameters.

The healthy group will eat 100 gr of Lettuce and 100 gr of biostimulated lettuce and will be collect plasma and urine samples after 15 days. Each subject will be subjected to two venous blood samples taken at the beginning of the observation and at the end. The samples obtained will be transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the experimenters at the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Samples will be analyzed and compared for glucose, albumin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, uric acid, creatinine, AST, ALT, γ-GT, ALP, bilirubin, Ferritin, free Iron, transferrin, total proteins, Magnesium, Calcium, insulin, osteocalcin, hematocrit, hs-CRP, TSH, FT3, FT4. Bone metabolism (Osteocalcin, parathyroid hormone, CTX, Calcitonin), Vitamin D Calcium, Phosphate, Potassium, gastric hormones ( GIP, GLP1, GLP2, ghrelin, glucagon, PYY, CCK, leptin, resistin).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Caucasian
  * age: 18-90 years
  * currently injury free
  * Body mass index between 18.5 and 28 kg/m2

Exclusion Criteria:

Exclusion Criteria:

* bone fracture within the previous year
* use of medication or suffering from any condition known to affect bone, lipid, glucose, iron metabolism
* pregnancy
* breastfeeding
* current smokers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
hepatic metabolism | 15 days
  AST (aspartate transaminase) and ALT (Alanine aminotransferase) will be measured in serum will be assessed at baseline and after 15 days
iron metabolism | 15 days
  ferritin, transferrin, % saturation of transferrin will be measured in serum will be assessed at baseline and after 15 days
Lipid metabolism | 15 days
  triglycerides, HDL, LDL, cholesterol will be measured in serum will be assessed at baseline and after 15 days
Glucose metabolism | 15 days
  insulin, glucose will be measured in serum will be assessed at baseline and after 15 days
Gastrointestinal peptides and lipid hormones | 15 days
  Plasma concentrations of Gastrointestinal peptides (GLP-1, GLP-2, GIP, PYY, Ghrelin) and lipid hormones (leptin, resistin, adiponectin) will be assessed at baseline and after and after 15 days.
Serum bone remodelling markers | 15 days
  PTH, calcitonin, Vitamin D, Calcium, Phosphate, Potassium will be assessed at baseline and after and after 15 days.
Serum bone matabolism markers | 15 days
  bone resorption CTX and bone formation osteocalcin will be assessed at baseline and after 15 days.
body mass index (BMI) | 15 days
  Weight (Kg) Height (m) BMI (kg/m2)

SECONDARY OUTCOMES:
body composition | 15 days
  lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara Baldassano Professor, PhD, Principal Investigator — University of Palermo
Locations (1):
- NABbio, STEBICEF department, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No
Because is forbidden by the Italian Low

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT05971017/Prot_SAP_000.pdf